CLINICAL TRIAL: NCT02661737
Title: A Multi-center, Prospective and Observational Study to Evaluate Long-term Safety and Biodegradability of Modified Sodium Hyaluronate Gel (YVOIRE Volume s) Injected for Correction of Nasolabial Folds
Brief Title: Observational Study to Evaluate Long-term Safety and Biodegradability of YVOIRE Volume s
Status: Completed | Type: Observational
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-HAOS005
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-11

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- YVOIRE volume s: Treatment with YVOIRE volume s
  Interventions: Device: YVOIRE volume s

INTERVENTIONS:
Device: YVOIRE volume s

SUMMARY:
To evaluate long-term safety of YVOIRE volume s by incidence of adverse events including injection site local reactions and biodegradability.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose age is over 18 years old and under 65 years old
2. Subjects whose WSRS grade is equal or greater than 2
3. Subjects must be willing and able to provide written informed consent form
4. Subjects who are scheduled to be treated with YVOIRE volumes for facial tissue augmentation to correct the nasolabial folds

Exclusion Criteria:

1. Subjects who are sensitive to hyaluronic acid or any excipients of YVOIRE volume s
2. Subjects who have received permanent implantation (silicone, PAAG, PMMA, CaHA etc) on the nasolabial folds
3. Subjects who have received nonpermanent aesthetic treatments, such as botulinum toxin injection or filler on the nasolabial folds within 9 months before screening
4. Subjects who have received face lifting or plastic surgery on face within 9 months before screening
5. Subjects who have received laser therapy on the nasolabial folds, chemical peeling or peeling on face within 3 months before the screening
6. Subjects who have any skin diseases (including inflammation and skin cancer) or infectious diseases on the injection sites
7. Subjects who tend to have hypertrophic scars
8. Subjects with a history of streptococcal disease, severe allergy or anaphylaxis or bleeding disorders.
9. Women in pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject who receive hyaluronic acid filler into the nasolabial folds
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- YVOIRE Volume s: YVOIRE volume s
  YVOIRE volume s
Period: Overall Study
Arm/Group | YVOIRE Volume s
Started | 503
Completed | 469
Not Completed | 34

BASELINE CHARACTERISTICS:
Arm/Group | YVOIRE Volume s
Number analyzed (Participants) | 469
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.58 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 462
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 469
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Device-related Adverse Events
Time Frame: Until subject reaching total biodegradation criterion (WSRS change) ; an expected average of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | YVOIRE Volume s
Number analyzed (Participants) | 503
Participants | 3

ADVERSE EVENTS:
Time Frame: Until subject reaching total biodegradation criterion (WSRS change) ; an expected average of 2 years
Arm/Group | YVOIRE Volume s
All-Cause Mortality (participants affected / at risk) | 0/503
Serious Adverse Events (participants affected / at risk) | 20/503
Other Adverse Events (participants affected / at risk) | 115/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | YVOIRE Volume s (N=503)
Breast disease (Injury, poisoning and procedural complications) | 4
Others (General disorders) | 16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | YVOIRE Volume s (N=503)
Dermatitis (Skin and subcutaneous tissue disorders) | 38
Upper respiratory tract infection (Infections and infestations) | 77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT02661737/Prot_SAP_000.pdf